CLINICAL TRIAL: NCT06224491
Title: Relationship Between Stress and Anxiety Levels and Ratings of Accompanying Non-occupational Symptoms in Vojta's Comprehensive RL Response
Brief Title: Non Motoric Reactions in Vojta Reflex Locomotion
Acronym: VojtaRL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Tereza Nováková, Tereza Nováková, PhD., Physiotherapy Deparment, Faculty of Physical Education and Sport, Charles University, Czech Republic
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 122111PRG
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Locomotion Disorder, Neurologic
Keywords: reflex locomotion according to Vojta, stress
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: These are healthy adult women. The expected number of participants is 20-30. To participate in the study, participants must agree to participate voluntarily. Contraindications for participation include psychiatric illness, cancer, acute inflammatory diseases, and pregnancy. Persons with signs of acute illness or injury or in recovery from acute illness or injury will not be eligible for testing. Subjects who, like the investigators, are students at FTVS UK will be personally approached and selected by the principal investigators. No email or phone number contacts will be used.
Who Masked: Participant
Masking Description: The participant is not familiar with the order of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo tactile stimulation (Sham Comparator): From a standardized starting position for 10 minutes tactile contact in the area outside the description of reflex zones in reflex locomotion according to Vojta.
  Interventions: Other: Reflex locomotion according to Vojta
- Reflex locomotion zone stimulation (Experimental): From a standardized starting position tactile stimulation in the area of the zone in reflex locomotion according to Vojta for 10 minutes .
  Interventions: Other: Reflex locomotion according to Vojta

INTERVENTIONS:
Other: Reflex locomotion according to Vojta — Tactile stimulation according to Vojta´s reflex locomotion
  Other Names: Placebo tactile stimulation.

SUMMARY:
Monitoring of non-motor manifestations of reflex locomotion according to Professor Vojta in laboratory conditions on healthy woman probands.

DETAILED DESCRIPTION:
The accompanying non-local manifestations during a maximum of 20 minutes of pressure stimulation of the zones defined by the concept of Professor Vojta will be observed. We will also examine the possible correlation between the magnitude of the response to Vojta Reflex Locomotion (VRL) and the degree of stress and anxiety on the part of the study participants. Approximately 20-30 participants will take part in the research. Manual stimulation of defined zones will be performed by an experienced physiotherapist who has successfully completed a course in the Vojta method. A Trigno Wireless EMG System Delsys device will be used to measure electrical muscle activity. Kistler force plates and a pliance-x® sensing system pedobarography device will be used to measure changes in standing. The SP-10 Pocket Spirometer Gima and wireless ECG will be used to measure changes in breathing and circulation. In addition, the DASS-42 and POMS questionnaires will be used. The aim of the study is to clarify whether during manual pressure stimulation of the zones defined by the above concept there is a change in electrical muscle activity, specific activity of the autonomic nervous system and whether there is a different partial pressure distribution in standing after the stimulation. Last but not least, the aim of the study is also to determine a possible correlation between the response rate to VRL and the level of stress and anxiety on the part of the study participants. All probands will be familiarized with the experimental measurement procedure and will sign an informed consent form prior to the start of the experiment. Measurements will be taken in the kinesiology laboratory of Physiotherapy department.

ELIGIBILITY:
Inclusion Criteria:

These will be healthy adult women. The expected number of participants is 20-30. To participate in the study, participants must agree to participate voluntarily.

Exclusion Criteria:

Contraindications for participation include psychiatric illness, cancer, acute inflammatory diseases, and pregnancy. Persons with signs of acute illness or injury or in recovery from acute illness or injury will not be eligible for testing.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Non-motor responses during tactile stimulation in reflex locomotion according to Vojta | 10 minutes tactile stimulation
  The Trigno Wireless EMG System Delsys will be used to measure electrical muscle activity. The SP-10 Pocket Spirometer Gima and wireless ECG will be used to measure changes in breathing and circulation. In addition, the DASS-42 and POMS questionnaires will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Charvátová, PhD., Study Chair — Faculty of Physical Education and Sport Charles University
Locations (1):
- Faculty of Physical Education and Sport, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
According to the possibility to share raw anonymised data.